CLINICAL TRIAL: NCT05347745
Title: An Interventional, Prospective IVD Device Study for the Testing of DNA Extracted from Tumor Tissue Biopsy Samples from Patients with Colorectal Cancer (CRC) Who Have Previously Tested Positive for KRAS G12C Mutation Into the Amgen Phase III Clinical Trial (Protocol No 20190172) to Demonstrate Clinical Performance of the Therascreen® KRAS RGQ PCR Kit.
Brief Title: Therascreen® KRAS RGQ PCR Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMF-20-1839-1-001
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2022-04

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Performance Study Protocol for therascreen® KRAS RGQ PCR Kit (Other): The therascreen® KRAS RGQ PCR Kit is a real-time qualitative PCR assay used on the Rotor-Gene Q MDx (US) instrument for the detection of seven somatic mutations in the human KRAS oncogene, using DNA extracted from formalin-fixed, paraffin-embedded (FFPE), colorectal cancer (CRC) tissue
  Interventions: Diagnostic Test: therascreen® KRAS RGQ PCR Kit

INTERVENTIONS:
Diagnostic Test: therascreen® KRAS RGQ PCR Kit — Utilize a Clinical Trial Assay, the KRAS Kit, as a screening test in Phase 3 of Clinical Study (Protocol No. 20190172) in order to identify patients with CRC with KRAS G12C mutation positive tumors This will allow the clinical data from the study to be used to determine the drug-device efficacy to support future regulatory submissions for the device-drug combination.

SUMMARY:
An interventional, prospective IVD device study for the testing of DNA extracted from tumor tissue biopsy samples from patients with Colorectal Cancer (CRC) who have previously tested positive for the KRAS G12C mutation for potential inclusion into the Amgen Phase III clinical trial (Protocol No 20190172) to demonstrate clinical performance of the therascreen® KRAS RGQ PCR Kit

DETAILED DESCRIPTION:
This is an interventional, prospective clinical performance study protocol for the testing of DNA extracted from tumor tissue biopsy samples obtained from patients with CRC using the KRAS kit.

(RES, CNB are acceptable however (Fine needle aspiration (FNA), brushings, cell pellets from pleural effusion, bone biopsy and lavage samples are not acceptable.

Up to 200 patient tissue samples (from approximately 100 clinical trial sites), obtained in the Clinical Study (Protocol No. 20190172), will be tested using the KRAS Kit. The testing will be performed at the l device clinical testing sites, Q2 Solutions Laboratories in the two geographical locations: USA and UK.

The clinical study protocol (Protocol No. 20190172) requires an estimated total of 153 evaluable patient tissue biopsy samples to be tested. Approximately 200 patient biopsy samples are expected to be supplied to the test sites to reach this target.

The KRAS G12C mutation status of patients enrolling on the clinical trial is expected to be known prior to patient screening hence the relatively low estimate of screen failures. If existing local data are used for patient selection, the archival tumor sample is requested to be sent to the Test Site for confirmation of KRAS G12C status prior to enrollment. For the US (Site 001) and EU (Site 002) Test Sites a FFPE tissue block (preferred) and a copy of the de-identified pathology report is requested by the Test Site or a minimum of 9 - 20 unstained slides (4-5 µm) should be submitted during screening for prospective central confirmation.

If no remaining tumor tissue is available from the biopsy used for determining KRAS G12C status then an alternative archival tumor sample may be submitted to the Test Site. If this is unavailable or if there is insufficient quality of tumor sample, a new biopsy will need to be provided for central KRAS G12C confirmation.

The primary objective of the Amgen Clinical Study is to evaluate the progression free survival assessed by MODIFIED RECIST 1.1 criteria of Sotorasib (AMG 510) at 2 different dose levels as a combination therapy with panitumumab, compared to patients treated with investigators choice comparator (trifluridine and tipiracil or regorafenib) in patients using the Clinical Study Assay, therascreen®KRAS Kit to assess the presence of the KRAS G12C mutation in CRC, a key eligibility criteria.

The clinical data from the study will be used to determine the drug-device efficacy to support future regulatory submissions for the device-drug combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically documented metastatic colorectal cancer (CRC).
2. Patients identified for inclusion in the Amgen Clinical Study (Protocol No. 20190172) who have signed and dated a valid informed consent form.
3. Patients must provide an archival tumor sample or a fresh tumor biopsy at baseline if an appropriate archival sample is unavailable.
4. Local KRAS data must be available for patient selection.
5. An archival tumor sample or fresh tumor biopsy is required for central confirmation of KRAS G12C status prior to enrollment.
6. Patient samples must meet the following criteria:

   1. A formalin-fixed paraffin-embedded (FFPE) tissue block (preferred) along with a de-identified pathology report.
   2. If an FFPE tissue block is unavailable, a minimum of 9-20 unstained slides (4-5 μm) must be submitted during screening for prospective central confirmation.
   3. If remaining tumor tissue from the KRAS status biopsy is unavailable, an alternative archival tumor sample may be submitted.
   4. If an alternative archival sample is unavailable or of insufficient quality, a new biopsy must be provided for central KRAS G12C confirmation.

   Submitted slides must be prepared using positively charged glass slides and cut within the past five years.
7. Patient samples must have been collected using one of the following methods:

   1. Core needle biopsy (CNB)
   2. Surgical resection (RES)
   3. Lavage samples

Exclusion Criteria:

1. Patients who do not meet all eligibility criteria for the Amgen Clinical Study (Protocol No. 20190172).
2. Patients with samples collected using one of the following methods:

   1. Fine needle aspiration (FNA)
   2. Brushings
   3. Cell pellets from pleural effusion
   4. Bone biopsy

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
therascreen® KRAS RGQ PCR Kit | 5 business days
  Device study is to utilize a Clinical Trial Assay, the KRAS Kit, as a screening test in Phase 3 of Clinical Study (Protocol No. 20190172) in order to identify patients with CRC with KRAS G12C mutation positive tumors
The number of patients identified for enrollment into Amgen's Phase III clinical trial based on a KRAS G12C mutation detected test result. | 12 months
  The primary objective of this device clinical performance study was to screen patients and confirm eligibility for enrollment into Amgen Phase III trail based on the detection of a KRAS G12C biomarker. If patents met all other eligibility criteria and were found to be KRAS G12C positive, they may enroll in the clinical trial. The primary outcome measure is the proportion pf patients tested with the QIAGEN therascreen KRAS RGQ PCR Kit that were KRAS G12C positive.

CONTACTS AND LOCATIONS:
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No